CLINICAL TRIAL: NCT02882828
Title: Pharmacokinetic Assessment of Tacrolimus Exposure Before and After a Switch From Twice Daily Immediate-release (Prograf®) to Once-daily Prolonged Release Tacrolimus (Envarsus®)
Brief Title: PK Assessment of Tacrolimus Exposure Before and After a Switch From Twice Daily Immediate-release (Prograf®) to Once-daily Prolonged Release Tacrolimus (Envarsus®)
Acronym: ENVARSWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: I160015
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Allograft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS (dried blood spots) collection (Experimental): In this study, we make a switch from Prograf® to Envarsus®. Patients will be trained to collect their blood from a finger prick on filter paper. DBS will be done at home, collected on filter paper and mailed by the patients to a centralized laboratory (Department of Pharmacology, Toxicology and Pharmacovigilance at Limoges University Hospital), where tacrolimus concentration will be determined by HPLC-MS/MS
  Interventions: Drug: switched from Prograf® to Envarsus®

INTERVENTIONS:
Drug: switched from Prograf® to Envarsus®

SUMMARY:
Tools have been developed in our unit to calculate the inter-dose AUC (Area Under Curve) of immunosuppressive drugs (ISD) based on a limited number of blood concentrations (i.e., blood samples) using Bayesian methods. Since 2005, we have implemented these tools in an expert system and made them available to the transplant community through our very successful ISBA (Immunosuppressive drugs Bayesian dose Adjustment) website.

Briefly, we first need to develop a population pharmacokinetic model using rich pharmacokinetic (PK) profiles (about 10 samples per patient over the dosing interval). The model developed can then be used for inference of ISD PK parameters in new patients using Bayesian estimation. Bayes' theorem is based on conditional probability: individual PK parameters are estimated based on the known PK parameters in the population (mean and distribution), given the dose and concentrations observed in a patient. Our previous studies have shown that a limited sampling strategy (LSS) based on 3 samples collected within the first 3 hours after drug intake can estimate adequately the interdose AUC of ISD. In the present study, the AUC0-24h and the recommended dose will be calculated using Bayesian estimators previously developed using PK data from the clinical trials run by Veloxis, and proposed to the clinicians via a dedicated website comparable with ISBA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 year-old) male and female patients
2. Recipient of a single kidney or liver allograft
3. Patient transplanted for more than 2 weeks and less than 1 year at enrolment
4. Patient with stable Prograf® dose, defined by the following criteria:

   * Criterion 1: unchanged Prograf® dose for at least one week; if not, apply criterion #2
   * Criterion 2: unchanged Prograf® dose since the last two therapeutic drug monitorings (TDM)
5. Patient for whom the decision is made to switch from Prograf® to Envarsus®
6. Written informed consent obtained prior to any study-related procedure
7. Patient with tacrolimus C0 between 4 and 12 µg/L at V1
8. Patient with hematocrit > 27% at V1

Exclusion Criteria:

1. Patient presenting any contra-indication to tacrolimus according to the summary of product characteristics (SmPC) of Envarsus®
2. Recipient of any transplanted organ other than kidney or liver
3. Patient treated by Prograf® for less than 7 days at enrolment
4. Patient previously treated by any other investigational agent if it is not stopped at least 7 days prior to enrolment
5. Pregnant or lactating woman (based on declaration)
6. Patient under judicial protection
7. Patient incapable of understanding the purposes and risks of the study, who cannot give written informed consent, or who are unwilling to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-10; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Difference between the post-switch tacrolimus steady-state AUC0-24h (V4) and the pre-switch AUC0-24h (V2). | 3 days
  The tacrolimus AUC0-24h at V2 (patient on Prograf®) will be calculated by summing the morning and the evening tacrolimus AUC0-12h.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - University Hospital of Amiens, Amiens
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Lille, Lille
  - Limoges Hospital, Limoges
  - AP-HP, Paris
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Reims, Reims
  - University Hospital of Rouen, Rouen
  - University Hospital of Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monchaud C, Woillard JB, Crepin S, Tafzi N, Micallef L, Rerolle JP, Dharancy S, Conti F, Choukroun G, Thierry A, Buchler M, Salame E, Garrouste C, Duvoux C, Colosio C, Merville P, Anglicheau D, Etienne I, Saliba F, Mariat C, Debette-Gratien M, Marquet P. Tacrolimus Exposure Before and After a Switch From Twice-Daily Immediate-Release to Once-Daily Prolonged Release Tacrolimus: The ENVARSWITCH Study. Transpl Int. 2023 Aug 1;36:11366. doi: 10.3389/ti.2023.11366. eCollection 2023. PMID 37588007